CLINICAL TRIAL: NCT00721539
Title: A Pilot Study Assessing Transoral Robotic Surgery (TORS) For Oral And Laryngopharyngeal Benign And Malignant Lesions Using The da Vinci® Robotic Surgical System
Brief Title: Assessing the da Vinci® Robotic Surgical System for Surgery of the Upper Aerodigestive Tract
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low Accrual
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Edward J. Damrose, Associate Professor of Otolaryngology, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: ENT0026; SU-07152008-1258 (Other: Stanford University)
Record Dates: First submitted 2008-07-22; First posted 2008-07-24 (Estimated); Results first posted 2016-11-03 (Estimated); Last update posted 2016-11-03 (Estimated); Status verified 2016-11

CONDITIONS: Hypopharyngeal Neoplasms; Laryngeal Neoplasms; Head and Neck Cancers
MeSH Terms: conditions — Hypopharyngeal Neoplasms; Laryngeal Neoplasms; Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Transoral Robotic Surgery (Other): Pilot study; single arm - use of da Vinci Surgical Robot Platform to access neoplastic disease of the upper aerodigestive tract.
  Interventions: Device: da Vinci Surgical Robot Platform; Procedure: Transoral Robotic Surgery

INTERVENTIONS:
Device: da Vinci Surgical Robot Platform — daVinci Surgical Robot Platform is a surgical device that enhances transoral access to the upper aerodigestive tract through miniaturization of endoscopes and micromanipulators that can be introduced through the mouth.
Procedure: Transoral Robotic Surgery — Eligible patients will undergo transoral treatment of neoplastic disease of the upper aerodigestive tract using the daVinci Surgical Robot Platform as opposed to traditional (TOL - transoral laser; TEC - transoral electrocautery) methods.

SUMMARY:
To assess the use of the da Vinci® Robotic Surgical System (Intuitive Surgical, Inc., Sunnyvale, CA) in transoral surgeries in patients with benign and malignant lesions of the oral cavity and laryngopharynx.

DETAILED DESCRIPTION:
In the past two decades the interest in minimally invasive techniques for transoral treatment of head and neck benign and malignant lesions has been growing due to the decreased morbidity of transoral approaches, and some surgeons have been moving away from traditional open resections. Transoral resection of neoplasms of the upper aerodigestive, by its minimally invasive nature, may afford a shorter hospitalization and recovery time for patients when compared to those patients who undergo traditional "open" surgery. In surgery of the oropharynx, hypopharynx, and larynx, transoral endoscopic surgery can provide similar outcomes in terms of local control of disease when compared to open procedures, while improving time to restoration of oral intake and shortening time to tracheostomy decannulation. Therefore, in select patients, a transoral surgical approach may afford clear advantages over traditional open approaches. Current techniques, however, are limited by the inability to attain direct line of site exposure of the lesion. Use of robot-assisted technology as a means to overcome surgical limitations, to provide surgeons with improved dexterity and precision, and to couple advanced imaging techniques with three-dimensional depth perception, may allow for the completion of transoral surgical approaches in patients for whom conventional technology has been suboptimal.

The da Vinci® Robotic Surgical System (Intuitive Surgical, Inc., Sunnyvale, CA) is FDA-approved for use in a variety of laparoscopic, thoracoscopic, cardiac, and urologic surgical procedures. This protocol will assess the use of the da Vinci® Robotic Surgical System (Intuitive Surgical, Inc., Sunnyvale, CA) in transoral surgeries in patients with benign and malignant lesions of the oral cavity and laryngopharynx. Traditional endoscopic removal of tumors of the oropharynx and laryngopharynx is usually preferred to traditional open resection because of the decrease in morbidity and improved functional outcomes experienced by patients. The limiting step in these procedures has been exposure of, visualization of, and access to candidate tumors. The da Vinci surgical system offers the possibility of significant improvements in exposure, visualization and access to these candidate tumors with no added risk to patients. Overall this may significantly increase the number of patients who are candidates for endoscopic surgery. Alternative procedures will include traditional open surgical removal of tumors as well as traditional endoscopic removal of tumors using the microscope and CO2 laser. Open surgical approaches are reserved for patients who have large tumors unsuitable for endoscopic removal or in whom endoscopic visualization of the tumor is inadequate or impossible. The da Vinci surgical system would offer improved visualization of tumors that might otherwise be inaccessible to a traditional endoscopic approach.

Candidate patients will present with a neoplasm of the oropharynx, hypopharynx or larynx. Those patients assessed preoperatively to be candidates for transoral surgery (eg, Mallampati class I or II, normal range of neck motion, no trismus) will undergo surgery via a transoral approach to resect the tumor. This will require general anesthesia and may require postoperative hospitalization. If the tumor can be accessed, resection will proceed using the da Vinci robot. In whom the tumor cannot be accessed, resection will proceed via the conventional open approach. Pre and postoperative care will not be affected by this protocol, as it deals strictly with the manner in which the tumor is removed. Postoperative care and visits are standardized as to the nature of the tumor (eg, malignant tumors usually require follow-up visits every four to six weeks to monitor for tumor recurrence). Complications, blood loss, operative time, length of hospitalization, time to resumption of oral intake, time to decannulation, and overall local control rates will be assessed in the postoperative period.

ELIGIBILITY:
Inclusion Criteria:

* Patient or volunteer is 18 years of age or older
* Patients must have indication for diagnosis and/or therapy of diseases of the oropharynx, hypopharynx, and/or larynx.

Exclusion Criteria:

* unexplained fever and/or untreated
* active infection
* pregnancy
* anatomic parameters which preclude transoral surgery, such as:

  1. trismus
  2. limited range of neck motion
  3. poor dentition
  4. redundant hypopharyngeal or supraglottic tissue which would prevent adequate visualization of the tumor
* participation in a research protocol which precludes participation in other protocols

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2010-09; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward J. Damrose MD, FACS, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients recruited through tertiary care medical center specializing in head and neck cancer; enrollment dates 9/2010 to 9/2012.
Pre-assignment Details: Exclusion criteria include unexplained fever, active infection, pregnancy, anatomic parameters which preclude surgery including trismus, limited range of neck motion, poor dentition, and physical features such as redundant hypopharyngeal tissues which prevent adequate exposure of tumor.
Period: Overall Study
Arm/Group | Transoral Robotic Surgery
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Transoral Robotic Surgery
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 7
  >=65 years | 1
Age, Continuous [Mean (Full Range); unit: Years] | 41.5 [18 to 65]
Gender [Count of Participants; unit: Participants]
  Female | 2
  Male | 7
Region of Enrollment [Number; unit: participants] — Adult patients from a tertiary referral academic center
  participants
    United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Overall Complication Rate (Intraoperative and Postoperative)
Description: Complications encountered intraoperatively or up to six weeks postoperatively. This would include injury to patient, hemorrhage, lacerations, and readmission following surgery.
Time Frame: Six weeks
Population: Subjects enrolled in this pilot study.
Measure: Number; unit: Participants
Arm/Group | Transoral Robotic Surgery
Number analyzed (Participants) | 9
Participants | 0

2. Secondary Outcome: Feasibility Defined as Ability to Perform the Planned Diagnostic or Therapeutic Procedure
Time Frame: Six weeks
Population: Adult patients 18 years of age and over
Measure: Number; unit: Participants
Arm/Group | Transoral Robotic Surgery
Number analyzed (Participants) | 9
Participants | 9

3. Secondary Outcome: Average Blood Loss
Description: Blood lost during procedure
Time Frame: Duration of procedure up to two hours
Population: Participants
Measure: Mean (Full Range); unit: mL
Arm/Group | Transoral Robotic Surgery
Number analyzed (Participants) | 9
mL | 50 [0 to 150]

4. Secondary Outcome: Average Operative Time
Description: Average operative time in minutes
Time Frame: Up to four hours (240 minutes)
Population: Participants
Measure: Mean (Full Range); unit: Minutes
Arm/Group | Transoral Robotic Surgery
Number analyzed (Participants) | 9
Minutes | 112 [38 to 208]

ADVERSE EVENTS:
Time Frame: Six weeks from the surgical date for each subject
Arm/Group | Transoral Robotic Surgery
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 0/9

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed secondary to low accrual of subjects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No